CLINICAL TRIAL: NCT01601457
Title: A Single-centre, Randomised, Double-blind, Parallel Group, Placebo-controlled Trial Evaluating the Efficacy and Safety of Activated Recombinant Coagulation Factor VII (rFVIIa, NovoSeven®) in Patients With Major Fractures of Pelvis or Pelvis and Acetabulum Undergoing Repair Surgery
Brief Title: Activated Recombinant Human Factor VII in Pelvic-acetabular Fracture Reconstruction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F7ORTHO-1506
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activated recombinant human factor VII (Experimental)
  Interventions: Drug: activated recombinant human factor VII
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: activated recombinant human factor VII — 90 mcg/kg body weight administered intravenously as a slow, bolus injection after the patients had been anaesthetised and immediately before the first skin incision. A second dose was given if an intraoperative haemoglobin was less than 8.0 g/dl after salvaged red cells (RBC) had been re-transfused
  Arms: Activated recombinant human factor VII
Drug: placebo — Administered intravenously as a slow, bolus injection after the patients had been anaesthetised and immediately before the first skin incision. A second dose was given if an intraoperative haemoglobin was less than 8.0 g/dl after salvaged red cells (RBC) had been re-transfused
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the efficacy of activated recombinant human factor VIIgiven in conjunction with standard therapy in patients undergoing major orthopaedic surgery following traumatic pelvic or pelvic and acetabular fractures.

ELIGIBILITY:
Inclusion Criteria:

* Injury due to a blunt or penetrating trauma causing pelvic or pelvic and acetabular fracture amenable to surgical reconstruction
* Scheduled for a semi-elective reconstruction surgery for fracture(s) of pelvis or pelvis and acetabulum, which was expected to be a "large" complex procedure with the potential of blood loss more than 50% of circulating blood volume

Exclusion Criteria:

* A history of thrombosis (deep vein thrombosis, pulmonary embolism, cerebral thrombosis)
* Patients with severe head injuries or an abnormal computed tomography (CT) scan of the head due to head injuries
* Body weight exceeding 135 kg
* Cardiac arrest following trauma and prior to surgery
* Known congenital bleeding disorders
* Known pregnancy or positive pregnancy test at enrolment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2002-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Total volume of perioperative blood loss

SECONDARY OUTCOMES:
Volumes of intraoperative and postoperative blood loss
Volume of blood transfused during the perioperative period
Vital signs
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, London, United Kingdom

REFERENCES:
- [Result] Raobaikady R, Redman J, Ball JA, Maloney G, Grounds RM. Use of activated recombinant coagulation factor VII in patients undergoing reconstruction surgery for traumatic fracture of pelvis or pelvis and acetabulum: a double-blind, randomized, placebo-controlled trial. Br J Anaesth. 2005 May;94(5):586-91. doi: 10.1093/bja/aei102. Epub 2005 Feb 25. PMID 15734783
- [Result] Hsia CC, Chin-Yee IH, McAlister VC. Use of recombinant activated factor VII in patients without hemophilia: a meta-analysis of randomized control trials. Ann Surg. 2008 Jul;248(1):61-8. doi: 10.1097/SLA.0b013e318176c4ec. PMID 18580208
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com